CLINICAL TRIAL: NCT02581111
Title: Randomized Placebo-controlled Trial of Intravenous Naloxone to Improve Oxygenation in Hypoxemic Lung-Eligible Brain-Dead Organ Donors
Brief Title: Naloxone for Optimizing Hypoxemia Of Lung Donors
Acronym: NO-HOLDS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Raj Dhar, Associate Professor of Neurology, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ODRC-001
Record Dates: First submitted 2015-10-01; First posted 2015-10-20 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Brain Death; Organ Donors; Lung Transplantation
MeSH Terms: conditions — Brain Death | interventions — Naloxone; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Naloxone (Experimental): Naloxone 8-mg IV given once after baseline ABG
  Interventions: Drug: Naloxone
- Placebo (Sham Comparator): Equivalent volume of saline given once
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Naloxone — Naloxone 8-mg IV bolus
  Other Names: Narcan
  Arms: Naloxone
Drug: Normal saline
  Other Names: saline
  Arms: Placebo

SUMMARY:
Brain-dead patients who provide authorization for organ donation will be randomized to naloxone or placebo if baseline arterial blood gas (ABG) after initiation of OPO (Organ Procurement Organization) management reveals hypoxemia, as defined by the ratio of partial pressure of oxygen in arterial blood (PaO2) to fraction of inspired oxygen (FiO2) below 300 mm Hg, unless they have already been ruled-out for lung recovery. Investigators aim to assess whether naloxone improves oxygenation prior to organ recovery more than placebo.

DETAILED DESCRIPTION:
Naloxone has been used by many OPOs for decades to improve the pulmonary status of brain-dead organ donors (based on anecdotal evidence and small uncontrolled studies). Its efficacy in this population has never been assessed in a controlled clinical trial. The rationale for its use appears to be that it blocks the increase in capillary permeability that occurs with herniation and brain death (as demonstrated in a single sheep study of herniation). Investigators aim to rigorously test this hypothesis in a randomized placebo-controlled trial in brain-dead organ donors who have baseline hypoxemia. The primary outcome will be the acute change in oxygenation (on first follow-up ABG after naloxone as well as the final ABG prior to organ recovery). Investigators will also assess whether treatment results in more lungs being recovered and transplanted, after correcting for baseline variables such as age, blood group, smoking history, and cause of death. This study will be performed under the auspices of the Organ Donation Research Consortium and be carried out by multiple OPOs across the country. Naloxone or blinded placebo (identical syringe filled with saline) will be given after the baseline ABG shows hypoxemia (PFR - PaO2 divided by FiO2, on positive end-expiratory pressure [PEEP] of 5 and usually 100% FiO2). Naloxone and placebo will both be co-administered with a neuromuscular blocking agent (e.g. vecuronium, per center protocol) to obviate any increase in spinal reflex movements that may be potentiated by naloxone treatment. All other protocols for organ donor management should be maintained at each OPO and no other study interventions are required. Transplant centers will be informed (through DonorNet) that the organ donor being considered for lung recovery has been enrolled in this blinded clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Brain-dead organ donor being managed by OPO (organ procurement organization)
* Lungs being considered for recovery and transplant
* Baseline ABG (after authorization) with P/F ratio < 300

Exclusion Criteria:

* No authorization for research
* Lungs already excluded for transplant (e.g. known chronic obstructive pulmonary disease [COPD], human immunodeficiency virus [HIV] infection)

Ages: 13 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-09-22 (Actual); Study Completion 2017-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajat Dhar, MD, Principal Investigator — Washington University School of Medicine
Locations (4):
- United States (4):
  - Donor Alliance, Denver, Colorado
  - Louisiana Organ Procurement Agency, Metairie, Louisiana
  - Mid-America Transplant Services, St Louis, Missouri
  - Lifeline of Ohio, Columbus, Ohio

REFERENCES:
- [Result] Dhar R, Stahlschmidt E, Paramesh A, Marklin G. A Randomized Controlled Trial of Naloxone for Optimization of Hypoxemia in Lung Donors After Brain Death. Transplantation. 2019 Jul;103(7):1433-1438. doi: 10.1097/TP.0000000000002511. PMID 30399122

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Equivalent volume of saline given once
  Normal saline
Period: Overall Study
Arm/Group | Naloxone | Placebo
Started | 98 | 101
Completed | 96 | 94
Not Completed | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naloxone | Placebo | Total
Number analyzed (Participants) | 98 | 101 | 199
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (13) | 36.8 (13) | 37 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 50 | 90
  Male | 58 | 51 | 109
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 13 | 18
  Not Hispanic or Latino | 87 | 83 | 170
  Unknown or Not Reported | 6 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 20 | 35
  White | 77 | 76 | 153
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  United States | 98 | 101 | 199

OUTCOME MEASURES:

1. Primary Outcome: Change in Oxygenation (P/F Ratio) From Baseline to Final Pre-recovery Arterial Blood Gas (ABG)
Description: Change in ratio of partial pressure of oxygen in arterial blood (PaO2) to fraction of inspired oxygen (FiO2) from final ABG performed before organ recovery compared to baseline ABG
Time Frame: Baseline and at time of organ recovery, within 72 hours
Measure: Median (Inter-Quartile Range); unit: mm Hg
Arm/Group | Naloxone | Placebo
Number analyzed (Participants) | 96 | 94
mm Hg | 81 [19 to 176] | 80 [-13 to 189]

2. Secondary Outcome: Number of Participants Who Had Lungs Transplanted
Description: Whether one or both lungs were transplanted from this organ donor (dichotomized)
Time Frame: At time of organ recovery (within 72 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Naloxone | Placebo
Number analyzed (Participants) | 98 | 101
Participants | 19 | 19

3. Secondary Outcome: Acute Change in Oxygenation (P/F Ratio)
Description: Change in PaO2:FiO2 ratio from ABG at 4-6 hours after randomization compared to baseline prior to randomization
Time Frame: Baseline and ABG at 4-6 hours after intervention
Measure: Median (Inter-Quartile Range); unit: mm Hg
Arm/Group | Naloxone | Placebo
Number analyzed (Participants) | 98 | 101
mm Hg | 71 [-9 to 129] | 33 [-12 to 111]

ADVERSE EVENTS:
Time Frame: Till organ recovery (maximum of three days)
Arm/Group | Naloxone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/101
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/101
Other Adverse Events (participants affected / at risk) | 0/98 | 0/101

LIMITATIONS AND CAVEATS:
10 subjects were enrolled despite baseline PaO2:FiO2 ratio above 300 (i.e. protocol violations)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-08-14): https://cdn.clinicaltrials.gov/large-docs/11/NCT02581111/Prot_000.pdf
  • Statistical Analysis Plan (2015-08-14): https://cdn.clinicaltrials.gov/large-docs/11/NCT02581111/SAP_001.pdf